CLINICAL TRIAL: NCT02065713
Title: A Multicentre, Randomized, Double-blind, Parallel-group Study To Compare The Efficacy Of Golimumab In Combination With Methotrexate (MTX) Versus MTX Monotherapy, In Improving Dactylitis And Enthesitis, In MTX Naïve Psoriatic Arthritis Patients.
Brief Title: Efficacy of Golimumab in Combination With Methotrexate (MTX) Versus MTX Monotherapy, in Improving Dactylitis, in MTX naïve Psoriatic Arthritis Patients
Acronym: GO-DACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Medicina Molecular João Lobo Antunes (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Elsa Vieira de Sousa, MD, Instituto de Medicina Molecular João Lobo Antunes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMM-50307
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis, dactylitis, enthesitis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — golimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Golimumab in combination with methotrexate (Experimental): Golimumab 50mg, subcutaneous, once monthly, for 24 weeks, in combination with MTX.
  MTX started at 15mg/weekly at baseline, increased to 20mg/weekly at week 4 and to 25mg/weekly at week 8, maintaining the dose of 25mg/weekly throughout the trial period of 24 weeks, except in case of intolerance or toxicity
  Interventions: Drug: Golimumab; Drug: Methotrexate
- Placebo in combination with methotrexate (Active Comparator): MTX started at 15mg/weekly at baseline, increased to 20mg/weekly at week 4 and to 25mg/weekly at week 8, maintaining the dose of 25mg/weekly throughout the trial period of 24 weeks, except in case of intolerance or toxicity.
  Interventions: Drug: Methotrexate; Drug: Placebo

INTERVENTIONS:
Drug: Golimumab — Prefilled syringe with golimumab 50mg (Simponi®) administrated subcutaneously, once monthly, for 24 weeks.
  Arms: Golimumab in combination with methotrexate
Drug: Methotrexate — MTX started at 15mg/weekly at baseline, increased to 20mg/weekly at week 4 and to 25mg/weekly at week 8, maintaining the dose of 25mg/weekly throughout the trial period of 24 weeks, except in case of intolerance or toxicity
Drug: Placebo — The prefilled syringe with placebo will be administrated subcutaneously, once monthly, for 24 weeks.
  Arms: Placebo in combination with methotrexate

SUMMARY:
Dactylitis is a poor prognostic factor in psoriatic arthritis (PsA) patients. The efficacy of synthetic or biologic disease modifying anti-rheumatic drugs (DMARDs) on dactylitis has not been previously studied in randomized controlled trials as a primary endpoint.

In this investigator initiated clinical trial the investigators aim to test the hypothesis that the combination therapy of golimumab and methotrexate (MTX) will result in a significant improvement of dactylitis in comparison with MTX monotherapy, in MTX naïve psoriatic arthritis patients, at week 24. Similarly the efficacy on enthesitis, peripheral and axial involvement, skin and nail psoriasis, inflammation and damage of the feet and hands assessed by magnetic resonance imaging (MRI), composite indexes of disease activity, remission, function and quality of life will be determined.

This is a national multicentre, interventional, double-blinded, placebo-controlled, parallel design trial. 136 patients with active dactylitis, refractory to at least two systemic non-steroidal anti-inflammatory drugs (NSAIDs), at optimal dosage, for 3 months will be included and centrally randomized to golimumab in combination with MTX versus MTX monotherapy, in a 1:1 ratio. The study duration will be 24 weeks.

The investigators expect the results from this trial will contribute to a better definition of the treatment algorithm of PsA patients with dactylitis.

ELIGIBILITY:
Inclusion Criteria:

Each subject must be/have…..

* Able and willing to give written informed consent and comply with the requirements of the study protocol.
* Age ≥ 18 years old, at baseline. A subject may be of both gender and any race/ethnicity.
* PsA diagnosis according to Classification of Psoriatic Arthritis (CASPAR) criteria, established at least 3 months prior to screening.
* Active psoriatic arthritis, at the time of entry into the study, defined by:

  ≥1 tender dactylitis, refractory to at least two systemic NSAIDs, at optimal dosage, for 3 months and at least one other site of active inflammation (peripheral joints, enthesis, spine, skin or nails).
* Naïve to MTX therapy.
* Patients can have been previously treated with synthetic DMARDs (except MTX) or corticosteroids but must have withdrawn according to the following schedules:

  * All synthetic DMARDs and oral corticosteroids withdrawn at least two weeks prior to screening or 5 half lives according, to what is longer, except for leflunomide.
  * leflunomide ≥ 12 weeks or ≥ 2 weeks after standard cholestyramine or activated charcoal washout.
  * Up to a maximum of two local corticosteroids injection are allowed, administrated, at least four weeks prior to screening (indication for local corticoids injection is dependent on expert opinion decision).
  * NSAIDs (up to the maximum recommend dose) if the dose has been stable for at least 4 weeks prior to baseline and the patient is expected to remain on the baseline dose for the 6 months of the study.
* Female subjects or male subjects and his female sexual partner of childbearing potential must agree to use a medically accepted method of contraception prior to enrollment, while receiving protocol-specified medication and for 6 months after stopping the medication.

  * Medically accepted methods of contraception include condoms (male or female) with a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device (IUD), inert or copper containing IUD, hormone-releasing IUD, systemic hormonal contraceptive, and surgical sterilization (eg, hysterectomy or tubal ligation). Other methods may be used as required by local legislation.
  * Postmenopausal women are not required to use contraception (postmenopausal is defined as at least 12 consecutive months without a spontaneous menses).

Exclusion Criteria:

A subject meeting any of the exclusion criteria listed below must be excluded from participating in the trial.

The subject has ….

* Known or suspected allergy to trial product or related products.
* Body weight > 100 Kg.
* Current chronic inflammatory autoimmune disease other than PsA that might confound the evaluations of safety and toxicity such as, but not limited to, ankylosing spondylitis, rheumatoid arthritis, tophaceous gout, reactive arthritis, pseudogout, arthropathy of inflammatory bowel disease, systemic erythematosus lupus, mixed connective tissue disease, scleroderma or variants, and polymyositis
* Active current infection or history of recurrent or chronic bacterial, viral, fungal, mycobacterial or other infections, including but not limited to tuberculosis and atypical mycobacterial disease, hepatitis B and C, HIV and herpes zoster.
* History of severe systemic bacterial, viral or fungal infections within the past 12 months prior to screening.
* Past or current malignancy with the exception of:

  * Adequately treated and cured basal cell carcinoma of the skin occurring more than 12 months prior to screening.
  * Other cancer with a complete response duration of > 5 years or any period of time longer than that, respectively for those malignancies which are considered as resolved after passing this duration of response.
* Any clinically significant medical condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the trial evaluations or patients safety and optimal participation in the trial such as, but not limited to:

  * Moderate to severe heart failure (New York Heart Association class III/IV)
  * Pre-existing central nervous system demyelinating disorders
  * Increased liver enzymes: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN).
* Female subject must not be breast-feeding.
* Female subject must not be pregnant or intending to become pregnant.
* Any contra-indications to perform MRI:

  * Patients who have a metal device affected by MRI
  * Allergy or other contraindications to an i.v. injection of gadolinium-diethylenetriamine pentaacetic acid
  * Claustrophobia sufficient to interfere with the patient undergoing the MRI scan.
* Previous treatment with tumor necrosis factor (TNF) blocking therapy or other biologic agents.
* Previous MTX therapy.
* Latent tuberculosis, in the absence of at least one month of isoniazid therapy, according to local guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Vieira de Sousa, MD, Principal Investigator — Instituto de Medicina Molecular João Lobo Antunes
Locations (1):
- Centro Académico de Medicina de Lisboa, Lisbon, Portugal

REFERENCES:
- [Derived] Vieira-Sousa E, Alves P, Rodrigues AM, Teixeira F, Tavares-Costa J, Bernardo A, Pimenta S, Pimentel-Santos FM, Gomes JL, Aguiar R, Pinto P, Videira T, Catita C, Santos H, Borges J, Sequeira G, Ribeiro C, Teixeira L, Avila-Ribeiro P, Martins FM, Canhao H, McInnes IB, Ribeiro RM, Fonseca JE. GO-DACT: a phase 3b randomised, double-blind, placebo-controlled trial of GOlimumab plus methotrexate (MTX) versus placebo plus MTX in improving DACTylitis in MTX-naive patients with psoriatic arthritis. Ann Rheum Dis. 2020 Apr;79(4):490-498. doi: 10.1136/annrheumdis-2019-216500. PMID 32193187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GO-DACT was a proof-of-concept multicentric, investigator-initiated trial conducted between August 2014 and June 2017, in 13 Rheumatology centres in Portugal.
Groups:
- Placebo in Combination With Methotrexate: Methotrexate (MTX) started at 15mg/weekly at baseline, increased to 20mg/weekly at week 4 and to 25mg/weekly at week 8, maintaining the dose of 25mg/weekly throughout the trial period of 24 weeks, except in case of intolerance or toxicity.
  Methotrexate: MTX started at 15mg/weekly at baseline, increased to 20mg/weekly at week 4 and to 25mg/weekly at week 8, maintaining the dose of 25mg/weekly throughout the trial period of 24 weeks, except in case of intolerance or toxicity
  Placebo: The prefilled syringe with placebo will be administrated subcutaneously, once monthly, for 24 weeks.
- Golimumab in Combination With Methotrexate: Golimumab 50mg, subcutaneous, once monthly, for 24 weeks, in combination with MTX.
  MTX started at 15mg/weekly at baseline, increased to 20mg/weekly at week 4 and to 25mg/weekly at week 8, maintaining the dose of 25mg/weekly throughout the trial period of 24 weeks, except in case of intolerance or toxicity
  Golimumab: Prefilled syringe with golimumab 50mg (Simponi®) administrated subcutaneously, once monthly, for 24 weeks.
  Methotrexate: MTX started at 15mg/weekly at baseline, increased to 20mg/weekly at week 4 and to 25mg/weekly at week 8, maintaining the dose of 25mg/weekly throughout the trial period of 24 weeks, except in case of intolerance or toxicity
Period: Overall Study
Arm/Group | Placebo in Combination With Methotrexate | Golimumab in Combination With Methotrexate
Started | 23 | 21
Completed | 22 | 20
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Golimumab in Combination With Methotrexate | Placebo in Combination With Methotrexate | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46.2 [34.9 to 50.4] | 44.1 [34.5 to 59.1] | 45.7 [34.8 to 54.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 17 | 20 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 22 | 42
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Portugal | 21 | 23 | 44
Dactylitis Severity Score (DSS) [Median (Inter-Quartile Range); unit: score on a scale] — Each digit with dactylitis was evaluated in a severity scale from 0 to 3 (0 = no dactylitis; 1 = mild dactylitis, 2 = moderate dactylitis, 3 = severe dactylitis). The total score is calculated as the sum of the individual digits dactylitis scores, ranging from a minimum 0 to a maximum of 60, with higher scores corresponding to worse severities.
  score on a scale | 6.0 [4.0 to 9.0] | 6.0 [4.5 to 8.0] | 6.0 [4.0 to 8.0]

OUTCOME MEASURES:

1. Primary Outcome: Dactylitis Severity Score (DSS)
Description: Changes from baseline in Dactylitis Severity Score at 24 weeks. Each digit with dactylitis was evaluated in a severity scale from 0 to 3 (0 = no dactylitis; 1 = mild dactylitis, 2 = moderate dactylitis, 3 = severe dactylitis). The total score is calculated as the sum of the individual digits dactylitis scores, ranging from a minimum 0 to a maximum of 60, with higher scores corresponding to worse severities.
Time Frame: From baseline to week 24
Population: An intention-to-treat analysis (ITT) was performed for the primary endpoint, applying the last observation carried forward method and including all randomly assigned patients who received at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: change of score on a scale
Arm/Group | Placebo in Combination With Methotrexate | Golimumab in Combination With Methotrexate
Number analyzed (Participants) | 23 | 21
change of score on a scale | -2 [-3.75 to -1.0] | -5 [-9.0 to -3.5]
Statistical Analysis 1: Comparison: Placebo in Combination With Methotrexate vs Golimumab in Combination With Methotrexate; Test type: Superiority; p = 0.026, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: For 32 weeks
Arm/Group | Placebo in Combination With Methotrexate | Golimumab in Combination With Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/21
Other Adverse Events (participants affected / at risk) | 14/23 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo in Combination With Methotrexate (N=23) | Golimumab in Combination With Methotrexate (N=21)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Worsening of polyarthritis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo in Combination With Methotrexate (N=23) | Golimumab in Combination With Methotrexate (N=21)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Lacrimal disorder (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (3)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza-like illness (General disorders) | 0 (0) | 1 (1)
Febrile infection (General disorders) | 0 (0) | 1 (1)
Cough (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Transaminases increased (Hepatobiliary disorders) | 4 (5) | 3 (3)
Alanine aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cutaneovisceral angiomatosis with thrombocytopenia (Immune system disorders) | 1 (1) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (2) | 0 (0)
Genital candidiasis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Viral rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Viral pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory tract infection viral (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Latent tuberculosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema eyelids (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Oral herpes (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Haematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 3 (3) | 0 (0)
Cervicalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gingivitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dental care (Surgical and medical procedures) | 0 (0) | 1 (1)
Herpetic gingivostomatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stomatitis aphthous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Molluscum contagiosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT02065713/Prot_SAP_000.pdf